CLINICAL TRIAL: NCT01111006
Title: The Effect of Electronic Cleansing Toilet System (Bidet) on Anal Resting Pressure in Normal Healthy Volunteers
Brief Title: The Effect of Electronic Cleansing Toilet System (Bidet) on Anal Resting Pressure
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Woongjin Coway Corporation (Unknown)
Responsible Party: Kyu Joo Park, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0620092310
Record Dates: First submitted 2010-04-04; First posted 2010-04-27 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Anorectal Physiology
Keywords: Electronic toilet; Bidet; Anorectal resting pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Bidet (electronic cleansing toilet system) — The volunteers underwent rectal examinations and baseline manometry at lateral decubitus position. Subjects were then placed on a toilet with Bidet attached and manometry catheter was inserted and fixed placing the channels of the catheter at the high pressure zone (HPZ) of the anal canal. Anorectal pressures were measured before and after using the Bidet under different water pressures (4, 8, 16, 20 gram force, gf), types of water stream (narrow vs. wide), and different temperatures (24oC vs. 38oC).
  Other Names: Bidet

SUMMARY:
The purpose of this study was to evaluate the effect of Bidet on anal resting pressure with regards to various flow rates and temperatures.

DETAILED DESCRIPTION:
Bidet is an electronic device spraying stream of the water for cleansing the anus and sometimes to aid defecation. It is widely used in Korea and Japan, with the flow rate (pressure) and temperature of water varying widely among the manufacturers. However, the effects of Bidet on anorectal function have not been studied in detail with regards to these variables.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer

Exclusion Criteria:

* anal disease pregnancy any medical disease that is necessary to treat psychosis

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The pressure before and after applying the bidet | after 1minute
  After the anal resting pressure was stabilized at sitting position, water stream of the bidet was applied to anus for 1 minute under various settings of different pressures (4, 8, 16, 20 gram force, gf), temperatures (24oC vs. 38oC), types of stream (narrow vs. wide) (Total time for experiment at individual subject was about two hours)

SECONDARY OUTCOMES:
The temperature of rectum | after 1minute
  The temperature probe was supposed to be placed in the rectum with manometry catheter and to prove the possibility of insertion of warm water into the rectum.

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Joo Park, MD, PhD, Principal Investigator — Department of Surgery, Seoul National University Hospital
Locations (1):
- Department of Surgery, Seoul National University Hospital, Seoul, Seoul, South Korea